CLINICAL TRIAL: NCT02727010
Title: Parenthood and Motherhood in Women With Motor Impairment and Disability Related to a Rare Disease
Brief Title: Motherhood With MOtor Impairment Due to MAlady (Rare Disease)
Acronym: MMOMA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Service d'Aide à la Parentalité des Personnes en Situation de Handicap (SAPPH) (Unknown)
Responsible Party: Sponsor
Other Study IDs: NI16003
Record Dates: First submitted 2016-03-29; First posted 2016-04-04 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2016-12

CONDITIONS: Disability Evaluation; Child of Impaired Parents
Keywords: Motor disability; Motor impairment; Pregnancy; Parenthood; Child psychology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- mothers with motor impairment due to a rare disease: 20 Women with motor impairment due to a rare disease
- mothers with motor impairment not related to a rare disease: controls, 20 women with motor impairment not related to a rare disease

SUMMARY:
Background Women with rare diseases resulting in motor disabilities wishing to become mother face a major challenge. The investigators hypothesize that provided with adequate support, they are able to achieve a successful pregnancy and to offer their child a safe family environment.

Methods To test this hypothesis, the investigators shall conduct a prospective observational prospective survey of a consecutive series of volunteer pregnant women or mothers of children less than 14 months, with motor impairment, participating in a program of parenting support developed in our institution.

Primary outcome: social environment, child development, mother-infant attachment, mother- infant interactions Secondary outcome: social and demographic characteristics, severity of motor impairment, associated impairment, perinatal morbidity for the mother and the infant (composite indicator), emotional status, and the needs expressed by women regarding the level of medical or social care.

Analysis The investigators shall describe the distribution of the primary outcome measurements in the subgroup of women with motor impairment related to a rare disease. The investigators shall compare this distribution to the expected distribution in the general population, and to that observed in women with motor impairment unrelated to a rare disease. The investigators shall also study primary outcome measurements as a function of the severity of maternal disability, of the mother's social characteristics and emotional status.

The investigators shall also describe the distribution the distribution of perinatal morbidity globally, and as a function of the potential explanatory variables mentioned above.

The investigators shall also report on the opinion of women regarding the support they were offered so far, and the support they declare they should benefit from.

DETAILED DESCRIPTION:
Background Women with motor disabilities have the same well-founded desire to become a mother as other women. Despite dedicated aids and adapted supportive measures, they face social blame from persons who believe they are not apt to provide adequate care to their children. When a rare disease caused the disability, planning to become a mother is even more critical, since most perinatal care providers are unfamiliar with the condition, and specialists of the disease are unfamiliar with pregnancy. Unsurprisingly, data on motherhood in women with rare diseases resulting in motor impairment are scarce.

The institutions of the investigators run a joint care program dedicated to future parents and parents with disabilities, namely:

* Hôpital Universitaire Pitié Salpêtrière- Charles Foix (assistance Publique Hôpitaux de Paris and Université Paris 6), providing a gynecological and perinatal unit with care programs adapted to women with disabilities, plus a number of reference centers for rare neurologic and muscular diseases including research and clinical care.
* Service d'Aide à la Parentalité des Personnes en Situation de Handicap (SAPPH, Fondation Hospitalière Sainte Marie) providing training and support to parenthood to persons with motor or sensory disabilities. This training program aims at recognizing parental capacities, and if necessary enhancing them by information, training, adapting the environment, or seeking extra human help.

The investigators felt the need to evaluate the outcome of our program, in terms of quality of infant environment, development, attachment, and interactions with their disabled mother. The investigators focused on parenthood in women with a rare disease resulting in motor impairment, a research field remaining largely unexplored so far.

Hypothesis Our hypothesis is that when provided with a specific care program, mothers with motor impairment due to a rare disease and their partners have the capacity to offer their children appropriate social environment and care, resulting in child development, mother-infant attachment, and mother- infant interactions being similar to what one would expect in women without motor impairment.

Objective Primary objective To describe social environment, child development, mother-infant attachment, mother- infant interactions, when the mother has motor impairment due du a rare disease.

Secondary objective

1. To describe maternal and perinatal outcome when the mother has motor impairment due du a rare disease
2. To explore a potential relation between the outcome criteria of the primary goal with

   * The severity of motor impairment
   * The causal disease
   * The personal history of the mother including her access to adapted care prior to pregnancy during pregnancy and post-partum
   * The social status of the family
   * The emotional status of the mother
3. To compare the distribution of primary goal outcome criteria in our study population to what is expected in the general population, when appropriate
4. To compare the distribution of primary goal outcome criteria in our study population to what we observed in women with motor impairment that does not result from a rare disease
5. To describe the needs expressed by women regarding medical care, psychological, social, and environmental support

Eligibility criteria Please see specific box

Outcome measurements (assessed at least once before the age of 14 months, see specific box) Primary outcome Child development /Infant attachment /Social environment /Mother infant interaction/ Child protection legal decisions if applicable Secondary outcome Demographic and social characteristics Disease or event causing impairment Obstetrical history Somatic and psychic events before, during pregnancy, and post-partum History of access to care Severity of impairment and handicap Maternal emotional status Needs expressed by women regarding medical care, psychological, social, and environmental support

Study design Pre inclusion: written and verbal information on the study to all women with motor impairment seeking care either at the Pitié Salpétrière Maternity unit or at the Service d'Aide à la Parentalité pour les Personnes en Situation de Handicap (SAPPH) Inclusion visit: During a planned training session, either pre natal or post natal Follow up visit: once of twice before the child is 14 months. A specific consent of both parents will be required for all outcome criteria concerning the infant.

Research visits will take place during usual visits of our parenthood support and training program.

Analysis The investigators shall describe the distribution of the primary outcome measurements in the subgroup of women with motor impairment related to a rare disease. The investigators shall compare this distribution to the expected distribution in the general population, and to that observed in women with motor impairment unrelated to a rare disease. The investigators shall also study primary outcome measurements as a function of the severity of maternal disability, of the mother's social characteristics and emotional status.

The investigators shall also describe the distribution the distribution of perinatal morbidity globally, and as a function of the potential explanatory variables mentioned above.

the investigators shall also report on the opinion of women regarding the support they were offered so far, and the support they declare they should benefit from.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 or older
* Either pregnant > 14 weeks, or mother of a child < 1 year
* With disability resulting from motor impairment
* Giving informed consent
* With social insurance

Exclusion Criteria:

* Know mental retardation
* Known psychiatric disorder
* Not fluent in French

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women or mothers to children < 14 months, with motor impairment, visiting the inclusion center and willing to participate in the study. Any motor impairment available, regardless of its cause.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Child development Mother infant attachment - Coding Interactive Behavior - Pirgas scale - Child protection legal decisions if applicable | At least once before the age of 14 months. May be repeated twice.
  Child development assessed by Brunet Lézine score: based on standardized examination of the infant by a trained child psychologist
Infant attachment | At least once before the age of 14 months. May be repeated twice.
  Infant attachment assessed by Guedenet and Fermanian ADBB scale: scale assessed by investigator
Social environment | At least once before the age of 14 months. May be repeated twice.
  Social environment assessed by Cutrona scale: self-administered questionnaire
Mother infant interaction | At least once before the age of 14 months. May be repeated twice.
  assessed by:
  * Coding Interactive Behavior: mother infant interaction filmed in a standardized fashion, and analyzed by trained psychologists blinded to the dyad's history.
  * Pirgas scale: clinical diagnosis regarding mother to infant interactions Child protection legal decisions : type of decision if applicable.

SECONDARY OUTCOMES:
Demographic and social characteristics | At lest once before the age of 14 months. May be repeated twice.
  Demographic and social characteristics, qualitative variables (Questionnaire administered by investigator)
Epices score of social deprivation | At lest once before the age of 14 months. May be repeated twice.
  Epices score of social deprivation (Self-administered questionnaire)
Disease or event causing impairment | At lest once before the age of 14 months. May be repeated twice.
  Disease or event causing impairment: preset qualitative variables (Questionnaire administered by investigator)
Obstetrical history | At lest once before the age of 14 months. May be repeated twice.
  Obstetrical history: preset qualitative variables (Questionnaire administered by investigator)
Somatic and psychic events before, during pregnancy, and post-partum (composite scores) | At lest once before the age of 14 months. May be repeated twice.
History of access to care | At lest once before the age of 14 months. May be repeated twice.
  History of access to care: standardized interview (Questionnaire administered by investigator)
Barthel score of capacity in everyday life | At lest once before the age of 14 months. May be repeated twice.
  Barthel score of capacity in everyday life (Self-administered questionnaire)
Ad hoc ordinal score based on the number of body parts with motor impairment and additional non-motor impairment | At lest once before the age of 14 months. May be repeated twice.
Maternal emotional status | At lest once before the age of 14 months. May be repeated twice.
  Assessed by STAI / EPDS scales (Self-administered questionnaire)
List of the needs expressed by women regarding medical care, psychological, social, and environmental support | At lest once before the age of 14 months. May be repeated twice.
  Assessed self-administered questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Drina Candilis, PhD, Principal Investigator — SAPPH
Locations (1):
- SAPPH, Paris, France

IPD SHARING:
Plan to Share IPD: No